CLINICAL TRIAL: NCT04111458
Title: A Phase I Open-label Dose Escalation Trial of BI 1701963 as Monotherapy and in Combination With Trametinib in Patients With KRAS Mutated Advanced or Metastatic Solid Tumours
Brief Title: A Study to Test Different Doses of BI 1701963 Alone and Combined With Trametinib in Patients With Different Types of Advanced Cancer (Solid Tumours With KRAS Mutation)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1432-0001; 2018-004757-24 (EudraCT Number)
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumors, KRAS Mutation; SOS1
Keywords: SOS1
MeSH Terms: interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 1701963 monotherapy (Experimental)
  Interventions: Drug: BI 1701963
- BI 1701963 + Trametinib (Experimental)
  Interventions: Drug: BI 1701963; Drug: Trametinib

INTERVENTIONS:
Drug: BI 1701963 — Tablet
Drug: Trametinib — Tablet
  Arms: BI 1701963 + Trametinib

SUMMARY:
This is a study in adults with advanced cancer (solid tumours) in whom previous chemotherapy was not successful. Only people who have a tumour with a KRAS mutation can participate in the study. A KRAS mutation makes cancer grow faster.

The study tests 2 medicines called BI 1701963 and trametinib. BI 1701963 prevents reactivation of KRAS. In this study, BI 1701963 is given to humans for the first time. Trametinib is an approved medicine (MEK inhibitor).

The purpose of this study is to find out the highest dose of BI 1701963 alone and in combination with trametinib the participants can tolerate. Another purpose is to check whether BI 1701963 in combination with trametinib is able to make tumours shrink.

Participants can stay in the study as long as they benefit from treatment and can tolerate it.

During this time, they get tablets of BI 1701963 and trametinib once daily. The doctors regularly monitor the size of the tumour. Doctors also regularly record any unwanted effects and check participants' health.

ELIGIBILITY:
Inclusion criteria:

All parts

* Previously-identified activating Kirsten rat sarcoma viral oncogene homologue (KRAS) mutation in tumour tissue or blood prior to screening
* At least one target lesion that can be measured per Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function
* Age ≥18 years of age, or over the legal age of consent as required by local legislation.
* Signed and dated written informed consent in accordance with GCP and local legislation prior to admission to the trial.
* Women of childbearing potential who are not surgically sterilized must have a negative serum pregnancy test completed during the Screening period
* Further inclusion criteria apply

Monotherapy and combination therapy dose escalation and monotherapy dose confirmation part

- Documented disease progression despite appropriate prior standard therapies or for whom no standard therapy exists for their tumour type and disease stage

Combination dose confirmation and expansion cohort

* Pathologically confirmed diagnosis of adenocarcinoma of the lung. Patients with mixed histology are eligible if adenocarcinoma is the predominant histology.
* Locally advanced stage IIIb or metastatic stage IV Non-small cell lung cancer (NSCLC)
* Patients must have received both chemotherapy and immunotherapy

Exclusion criteria:

All parts

* Previous anticancer chemotherapy within 3 weeks of the first administration of trial drug.
* Previous treatment with RAS, Mitogen-activated protein kinase (MAPK) or Son of sevenless 1 (SOS1) targeting agents
* Major surgery performed within 4 weeks prior to start of treatment
* Uncontrolled hypertension, congestive heart failure NYHA classification of ≥3, unstable angina or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to start of treatment
* Left ventricular ejection fraction (LVEF) <50 %
* Congenital long QT prolongation syndrome
* Mean resting corrected QT interval (QTcF) >470 msec
* Leptomeningeal carcinomatosis
* Presence or history of uncontrolled or symptomatic brain metastases
* Known pre-existing interstitial lung disease
* Known active hepatitis B infection (defined as presence of Hep B sAg and/or Hep B Deoxyribonucleic acid (DNA)), active hepatitis C infection (defined as presence of Hep C Ribonucleic acid (RNA))
* Active infectious disease
* Any history or presence of uncontrolled gastrointestinal disorders that could affect the intake and/or absorption of the trial drug
* History of retinal vein occlusion (RVO) or retinal pigment epithelial detachment (RPED)
* Further exclusion criteria apply

Combination part

- Hypersensitivity to any of the excipients listed in the current Summary of Product Characteristics (SmPC)/Package insert (PI) of trametinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose escalation (Part A) - Maximum tolerated dose (MTD) based on number of dose-limiting toxicities (DLTs) | 4 weeks
Dose confirmation (Part B) - Number of patients with DLTs during the on-treatment period | Up to 3 years
Dose confirmation (Part B) and expansion (Part C) - Objective response | Up to 3 years

SECONDARY OUTCOMES:
Dose escalation (Part A), confirmation (Part B) and expansion (Part C) - Pharmacokinetic parameters of BI 1701963: Cmax (maximum measured concentration of the analyte in plasma) | Up to 5 weeks
Dose escalation (Part A), confirmation (Part B) and expansion (Part C) - Pharmacokinetic parameters of BI 1701963: AUCτ (area under the concentration-time curve over a uniform dosing interval τ) | Up to 5 weeks
Dose escalation (Part A), confirmation (Part B) and expansion (Part C) - Pharmacokinetic parameters of trametinib: Cmax (maximum measured concentration of the analyte in plasma) | Up to 5 weeks
Dose escalation (Part A), confirmation (Part B) and expansion (Part C) - Pharmacokinetic parameters of trametinib: AUCτ (area under the concentration-time curve over a uniform dosing interval τ) | Up to 5 weeks
Dose confirmation (Part B) - Pharmacokinetic parameters of BI 1701963: Cmax (maximum measured concentration of the analyte in plasma) | Up to 5 weeks
Dose confirmation (Part B) - Pharmacokinetic parameters of BI 1701963: AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | Up to 5 weeks
Dose confirmation (Part B) - Pharmacokinetic parameters of midazolam: Cmax (maximum measured concentration of the analyte in plasma) | Up to 5 weeks
Dose confirmation (Part B) - Pharmacokinetic parameters of midazolam: AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | Up to 5 weeks
Dose confirmation (Part B) - Number of patients with Grade ≥3 treatment-related adverse events observed during the on-treatment period | Up to 3 years
Dose confirmation (Part B) and expansion (Part C) - Duration of Objective response (OR) | Up to 3 years
Dose confirmation (Part B) and expansion (Part C) - Tumour shrinkage (in millimetres) | Up to 3 years
Dose confirmation (Part B) and expansion (Part C) - Progression-free survival | 6 months
Dose confirmation (Part B) and expansion (Part C) - Number of patients with Grade ≥3 treatment-related adverse events observed during the on-treatment period | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Levine Cancer Institute, Charlotte, North Carolina
  - Sarah Cannon Research Institute-Nashville-48456, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Germany (2):
  - Universitätsklinikum Köln (AöR), Cologne
  - Universitätsklinikum Frankfurt, Frankfurt am Main
- Netherlands (2):
  - Erasmus Medisch Centrum-ROTTERDAM-50697, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor'
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com